CLINICAL TRIAL: NCT05747599
Title: Adapting and Testing a Behavioural Intervention to Prevent FASD and Adverse Infant Outcomes
Acronym: MaRISA+
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: Medical Research Council, South Africa (Other)
Responsible Party: Principal Investigator, Yukiko Washio, Principal Investigator, RTI International
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: EC025-11/2022
Record Dates: First submitted 2023-01-30; First posted 2023-02-28 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Maternal Behavior; Alcohol Drinking; Fetal Conditions
MeSH Terms: conditions — Alcohol Drinking | interventions — Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Contingent incentives on abstinence from alcohol, tobacco, and cannabis; Text-based support based on educational components
  Interventions: Behavioral: Intervention with contingent incentives and text-based support
- Usual Care (Active Comparator): Community treatment referrals
  Interventions: Behavioral: Intervention with contingent incentives and text-based support

INTERVENTIONS:
Behavioral: Intervention with contingent incentives and text-based support — Contingent incentives on abstinence from alcohol, tobacco, and cannabis; Text-based support based on educational components

SUMMARY:
South Africa (SA) has a long history of social and health disparities, resulting in the world's highest rate of fetal alcohol spectrum disorder (FASD; 111.1 per 1,000), where lifelong negative cognitive and physical effects result from prenatal alcohol exposure. FASD is completely preventable if women do not drink during pregnancy. Prenatal alcohol use frequently co-occurs with other substance use, especially tobacco and cannabis. The adverse effect on birth outcomes by alcohol and tobacco use together is worse than either substance alone. Recent evidence from animal models shows that prenatal exposure to both cannabinoids and alcohol potentiate the likelihood of alcohol-induced birth defects.

Data from Cape Metropole, SA, showed that all women who reported prenatal alcohol use also tested positive for tobacco use, with 25% also reporting cannabis use. Alcohol use while breastfeeding also occurs at a relatively high rate in SA. Despite tremendous health benefits from breastfeeding,maternal alcohol use while breastfeeding significantly compromises infant development. Contingency management (CM) has been efficacious in reducing prenatal cocaine, alcohol, and tobacco use in the United States (U.S.). The Women's Health CoOp (WHC) is an evidence-based brief intervention addressing women-focused syndemic issues and resulting disparities associated with substance and alcohol use. These evidence-based interventions need to be combined and adapted for addressing maternal polysubstance use and associated health and behavioral issues during pregnancy and lactation in SA. The Specific Aims are as follows: (1) R61 Aim 1- Conduct formative qualitative research with women who are pregnant or breastfeeding with a recent history of polysubstance use, clinic and community stakeholders, and an established Community Collaborative Board. (2) R61 Aim 2-Test feasibility, acceptability, and appropriateness of the adapted intervention with 48 women (24 pregnant and 24 breastfeeding) in Cape Metropole, SA. (3) R33 Aim 1-Examine the effectiveness of the adapted intervention (i.e., CM and text-based support with WHC educational components) in a 2-group randomized controlled trial with 184 women who are pregnant and follow up during pregnancy and 3 months postpartum. (4) R33 Aim 2-Examine the impact on gestational, birth, and infant outcomes. (5) R33 Aim 3-Track cost and conduct preliminary cost-effectiveness analyses.

ELIGIBILITY:
Inclusion Criteria:

For key informant interviews in R61 To be eligible, women must (1) 18 or older, (2) be pregnant or breastfeeding with less than 12 months postpartum, (3) report alcohol use , (4) report tobacco or cannabis use

For testing in R61,

1. be in the second trimester of pregnancy or breastfeeding with less than 3 months postpartum,
2. test positive in alcohol use by urinalysis (i.e., EtG),
3. test positive in tobacco or cannabis use by urinalysis (i.e., cotinine and THC),
4. be over 18 years old
5. have a negative HIV test,
6. not be eligible for PrEP
7. plan to complete antenatal care at the current clinic and remain in the area for at least 3 months
8. own a cell phone to receive text messages.

Exclusion Criteria:

- (1) women who report serious medical problems threatening their current pregnancy or current suicidal thoughts or attempts in the past month. These women will be provided necessary referrals.

(2) Women who participated in interviews.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yukiko Washio, PhD, Principal Investigator — RTI International
Locations (1):
- South African Medical Research Council, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: Yes
After the main findings are published, we welcome other researchers who want to analyze the data in other ways.
Supporting Information: Study Protocol, SAP, CSR

RESULTS

PARTICIPANT FLOW:
Groups:
- Contingent Incentives + Text-based Support: Contingent incentives on abstinence from alcohol, tobacco, and cannabis; Text-based support based on educational components
Period: Overall Study
Arm/Group | Contingent Incentives + Text-based Support
Started | 48
Completed | 45
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Contingent Incentives + Text-based Support: Contingent incentives on abstinence from alcohol, tobacco, and cannabis; Text-based support based on educational components
  Intervention with contingent incentives and text-based support: Contingent incentives on abstinence from alcohol, tobacco, and cannabis; Text-based support based on educational components
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 30 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mixed | 31
  Black | 17
Marital Status [Count of Participants; unit: Participants]
  Married | 9
  Living with a partner | 19
  Not living with a partner | 16
  Others | 4
Education [Count of Participants; unit: Participants]
  12 years or less | 44
  More than 12 years | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Urinalysis for Alcohol Metabolite (EtG)
Description: An alcohol metabolite (EtG) will be measured in urine samples. EtG can be detected in the urine up to 5 days after heavy drinking and up to 2 days after light drinking. The dipstick testing will have ≥300 ng/mL as a cutoff value.
Time Frame: 3-month postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Participants | 44

2. Primary Outcome: Number of Participants With Negative Urinalysis for Nicotine Metabolite (Cotinine)
Description: Biochemical verification of recent tobacco use in urine samples. A tobacco metabolite (cotinine) will be measured in urine samples. The metabolite can be detected up to 3-4 days after use. The dipstick testing will have ≥200 ng/mL as a cutoff value.
Time Frame: 3-month postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Participants | 18

3. Primary Outcome: Number of Participants With Negative Urinalysis for Cannabis Metabolite (THC)
Description: Biochemical verification of recent cannabis use in urine samples. A cannabis metabolite (THC) will be measured in urine samples. The metabolite can be detected up to 28 days after heavy use. The dipstick testing will have ≥50 ng/mL as a cutoff value.
Time Frame: 3-month postpartum
Measure: Count of Participants; unit: Participants
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Participants | 42

4. Primary Outcome: Number of Days in the Past 7-day Alcohol Use
Description: The number of days in the past 7 days that participants used alcohol.
Time Frame: 3-month postpartum
Measure: Mean (Standard Deviation); unit: Days in the past week alcohol use
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Days in the past week alcohol use | 0.2 (0.5)

5. Primary Outcome: Number of Days in the Past 7-day Tobacco Use
Description: The number of days in the past 7 days that participants used tobacco.
Time Frame: 3-month postpartum
Measure: Mean (Standard Deviation); unit: Days in the past week tobacco use
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Days in the past week tobacco use | 3 (3.4)

6. Primary Outcome: Number of Days in the Past 7-day Cannabis Use
Description: The number of days in the past 7 days that participants used cannabis.
Time Frame: 3-month postpartum
Measure: Mean (Standard Deviation); unit: Days in the past week cannabis use
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Days in the past week cannabis use | 0.4 (1.4)

7. Secondary Outcome: Number of Days in the Past 7-day Cannabis Use While Breastfeeding
Description: The number of days in the past 7 days that participants used cannabis while breastfeeding.
Time Frame: 3-month postpartum
Measure: Mean (Standard Deviation); unit: Days in the past week BF/Cannabis
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Days in the past week BF/Cannabis | 0.02 (0.1)

8. Secondary Outcome: Number of Days in the Past 7-day Tobacco Use While Breastfeeding
Description: The number of days in the past 7 days that participants used tobacco while breastfeeding.
Time Frame: 3-month postpartum
Measure: Mean (Standard Deviation); unit: Days in the past week BF/Smoking
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Days in the past week BF/Smoking | 2 (2.8)

9. Secondary Outcome: Number of Days in the Past 7-day Alcohol Use While Breastfeeding
Description: The number of days in the past 7 days that participants used alcohol while breastfeeding.
Time Frame: 3-month postpartum
Measure: Mean (Standard Deviation); unit: Days in the past week BF/Drinking
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 45
Days in the past week BF/Drinking | 0.1 (0.4)

10. Other Pre Specified Outcome: Birth Weight (g)
Description: birth weight of infants among participants who entered the study during pregnancy
Time Frame: at birth
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 23
grams | 2804 (407)

11. Other Pre Specified Outcome: Birth Length (cm)
Description: birth length of infants among participants who entered the study during pregnancy
Time Frame: at birth
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 22
cm | 48 (3)

12. Other Pre Specified Outcome: Gestational Age (Weeks)
Description: Gestational age of infants among participants who entered the study during pregnancy
Time Frame: at birth
Measure: Mean (Standard Deviation); unit: weeks
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 23
weeks | 38 (2)

13. Other Pre Specified Outcome: Head Circumference (cm)
Description: Head circumference of infants among participants who entered the study during pregnancy
Time Frame: at birth
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Contingent Incentives + Text-based Support
Number analyzed (Participants) | 22
cm | 33 (2)

ADVERSE EVENTS:
Time Frame: Approximately 6 months
Arm/Group | Intervention
All-Cause Mortality (participants affected / at risk) | 0/48
Serious Adverse Events (participants affected / at risk) | 2/48
Other Adverse Events (participants affected / at risk) | 2/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=48)
Infant death (Investigations) | 1 (1) — Unknown cause
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=48)
High blood pressure (Blood and lymphatic system disorders) | 1 (1)
Preterm labor (Pregnancy, puerperium and perinatal conditions) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-11): https://cdn.clinicaltrials.gov/large-docs/99/NCT05747599/Prot_SAP_ICF_000.pdf